CLINICAL TRIAL: NCT06530745
Title: Quintuple Intra-Articular Hyaluronic Acid (HA) Improves and Platelet-Rich Plasma (PRP) Does Not Affect Mandibular Mobility in Temporomandibular Joint (TMJ) Disorders: A Controlled Trial
Brief Title: PRP vs HA Intra-articular Injections in TMDs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital of the Ministry of Interior, Kielce, Poland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/2024/1
Record Dates: First submitted 2024-07-27; First posted 2024-07-31 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Temporomandibular Joint Disorders; Temporomandibular Joint Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Hyaluronic Acid; Injections

STUDY DESIGN:
Intervention Model Description: This study was designed as a two-arm equal-allocation clinical trial with a non-concurrent active treatment control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP receiving group (Experimental): Patients receiving platelet-rich plasma injections into temporomandibular joints.
  Interventions: Procedure: Platelet-rich plasma (PRP) injection
- HA receiving group (Active Comparator): Patients receiving hyaluronic acid injections into temporomandibular joints.
  Interventions: Procedure: Hyaluronic acid (HA) injection

INTERVENTIONS:
Procedure: Hyaluronic acid (HA) injection — 2% hyaluronic acid Synocrom Forte (Croma-Pharma GmbH, Leobendorf, Austria) injection
  Arms: HA receiving group
Procedure: Platelet-rich plasma (PRP) injection — PRP from peripheral venous blood of the elbow bend centrifuged at 160 revolutions per minute for 5 minutes with iFuge D06 (Neuation Technologies Pvt. Ltd, Gujarat, India) injection
  Arms: PRP receiving group

SUMMARY:
This clinical trial aims to compare the multidirectional mandibular mobility following the treatment of TMJ disorders with same-protocol intra-articular injections of PRP and HA. It is questioned whether there is direct clinical evidence of the superiority of PRP or HA in the injection treatment of TMJ disorders.

DETAILED DESCRIPTION:
This study was designed as a two-arm equal-allocation clinical trial with a non-concurrent active treatment control. The study group consisted of consecutive patients receiving PRP injections into the TMJ cavities. The control group consisted of the same number of patients who received HA according to the same protocol. Controls were recruited consecutively, men and women separately, to maintain a consistent male-to-female ratio. The main condition for recruitment was the diagnosis of TMJ pain by a specialist in orthodontics or dental prosthetics and, on this basis, a referral for injection treatment. TMJ pain was diagnosed under the ICOP 2020 guidelines. The treatment was performed at the Maxillofacial Surgery Clinic in Kielce, Poland. The study group received PRP from peripheral venous blood of the elbow bend centrifuged at 160 revolutions per minute for 5 minutes with iFuge D06 (Neuation Technologies Pvt. Ltd, Gujarat, India). The control group received 2% hyaluronic acid Synocrom Forte (Croma-Pharma GmbH, Leobendorf, Austria). In both groups, 0.4 mL of the solution was injected per joint.

ELIGIBILITY:
Inclusion Criteria:

* ICOP 2020 diagnosis of TMJ pain;
* informed consent to participate in the study;
* the possibility of discontinuing the current treatment of the temporomandibular joints;
* generally accepted indications for injection therapy.

Exclusion Criteria:

* active cancer;
* hematopoietic system disease or bleeding diathesis;
* temporomandibular joint prosthesis;
* temporomandibular joint ankylosis;
* skin disease of the preauricular area of the affected side.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Mandibular abduction | 0 - 6 months
  Range of mandibular abduction between anthropometric points Incision superius (Is) and Incision inferius (Ii)
Mandibular protrusion | 0 - 6 months
  Range of mandibular abduction between anthropometric points Incision superius (Is) and Incision inferius (Ii)
Mandibular right movement | 0 - 6 months
  Range of mandibular abduction between anthropometric points Incision superius (Is) and Incision inferius (Ii)
Mandibular left movement | 0 - 6 months
  Range of mandibular abduction between anthropometric points Incision superius (Is) and Incision inferius (Ii)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Sikora, dr hab., Study Chair — Hospital of the Ministry of Interior, Wojska Polskiego 51, 25-375 Kielce, Poland
Locations (1):
- Department of Maxillofacial Surgery, Kielce, Poland

IPD SHARING:
Plan to Share IPD: No